CLINICAL TRIAL: NCT00620958
Title: Parent Mediation of Child Anxiety CBT Outcome
Brief Title: Cognitive Behavioral Therapy With Parental Involvement for Treating Children With Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Wendy Silverman, Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH079943 (NIH); R01MH079943 (NIH); DSIR 84-CTS; 1R01MH079943-01A1 (NIH)
Record Dates: First submitted 2008-02-20; First posted 2008-02-22 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Anxiety Disorders
Keywords: Mediation; Outcome; CBT; Child Anxiety Intervention
MeSH Terms: conditions — Anxiety Disorders; Negotiating | interventions — Eukaryotic Initiation Factor-3

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive individual cognitive behavioral therapy with parent reinforcement training.
  Interventions: Behavioral: Parent reinforcement training (PRT1) With Individual Cognitive Behavioral Therapy (ICBT)
- 2 (Experimental): Participants will receive individual cognitive behavioral therapy with parent relationship training.
  Interventions: Behavioral: Parent relationship training (PRT2) With Individual Cognitive Behavioral Therapy (ICBT)
- 3 (Active Comparator): Participants will receive individual cognitive behavioral therapy alone.
  Interventions: Behavioral: Individual cognitive behavioral therapy (ICBT)

INTERVENTIONS:
Behavioral: Individual cognitive behavioral therapy (ICBT) — ICBT will include 12 to 14 sessions during which child participants will learn how to change anxious and fearful thoughts and to deal with feared objects and events.
  Other Names: CBT
  Arms: 3
Behavioral: Parent relationship training (PRT2) With Individual Cognitive Behavioral Therapy (ICBT) — Parent relationship training will teach the parent ways to communicate with the child and to solve problems to help discourage child avoidant behaviors. ICBT will include 12 to 14 sessions during which child participants will learn how to change anxious and fearful thoughts and to deal with feared objects and events.
  Arms: 2
Behavioral: Parent reinforcement training (PRT1) With Individual Cognitive Behavioral Therapy (ICBT) — Parent reinforcement training will teach the parent strategies for managing the child's behavior through the use of positive rewards and positive parental behaviors to help discourage child avoidant behaviors. ICBT will include 12 to 14 sessions during which child participants will learn how to change anxious and fearful thoughts and to deal with feared objects and events.
  Arms: 1

SUMMARY:
This study will compare the effectiveness of individual cognitive behavioral therapy with two distinct types of parent involvement versus individual cognitive behavioral therapy without parent involvement in treating children with anxiety disorders. Hypothesized mediator of change for eac of the two parent treatment conditions also will be evaluated

DETAILED DESCRIPTION:
Anxiety disorders are among the most common emotional, behavioral, and mental disorders in children, affecting an estimated 1 out of every 10 children and adolescents. Symptoms of anxiety disorders include an excessive sense of worry, stress, and fear; headache; nausea; and impaired learning and concentration. If left untreated, anxiety disorders can lead to difficulties with school and relationships, substance abuse, and the persistence of anxiety problems into adulthood. Individual cognitive behavioral therapy (ICBT), in which children learn to cope with fears through behavior and thought modification, has been an effective form of treatment for children with anxiety disorders. Studies have indicated that ICBT involving children and parents may be more effective than ICBT involving only children for improving anxiety levels and long-term recovery rates. This study will compare the effectiveness of ICBT with either parent reinforcement training or parent relationship training versus ICBT without parent involvement in treating children with anxiety disorders.

Participation in this study will last 15 months, with 3 months of treatment and 12 months of follow-up. Both parent and child participants will first undergo initial assessments that will include psychological questionnaires; a video-taped child-parent interaction session; and interviews about behaviors, psychological functioning, and problem situations. Participants will then be assigned randomly to one of three treatment groups: ICBT, ICBT with parent reinforcement training (PRT1), or ICBT with parent relationship training (PRT2). All participants will attend between 12 and 14 weekly treatment sessions, lasting 60 minutes each. During all sessions, child participants will learn how to change anxious and fearful thoughts and to deal with feared objects and events. ICBT PRT1 and ICBT PRT2 sessions will also involve the parent and child working together. ICBT PRT1 will specifically teach the parent strategies for managing the child's behavior through the use of positive rewards and positive parental behaviors to help discourage child avoidant behaviors. ICBT PRT2 will specifically teach the parent ways to communicate with the child and to solve problems to help discourage child avoidant behaviors.

All participants will be asked to complete questionnaires throughout treatment, upon completion of treatment, and 6 months after the end of treatment. Three and 9 months after the end of treatment, participants will undergo a 15-minute telephone assessment to evaluate how the child participant has been doing. The final assessment will occur 12 months after the end of treatment and will include repeat interviews and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for a primary diagnosis of an anxiety disorder, including generalized anxiety disorder (GAD), social phobia (SOP), and social anxiety disorder (SAD), as confirmed by ADIS C/P
* Receives a mean score of 4 or greater on the Clinician's Rating Scale of Severity (CSR)
* Willing to stop all other child psychosocial treatment upon study entry
* Comorbid attention deficit hyperactivity disorder (ADHD) and depressive disorders with CSR scores less than 4 are acceptable if treated and stable
* Tics or aggression/impulse control problems with minimal or no impairment are acceptable if treated and stable
* If taking medication, on stable medication treatment for comorbid ADHD, major depressive disorder, tics, or aggression/impulse control
* Agreement of parents or guardians to participate in the child participant's treatment
* Child living with a primary caregiver who has known the child well for at least 6 months and who is legally able to give consent for the child's participation

Exclusion Criteria:

* Meets as a primary diagnosis any Axis I DSM-IV disorder other than GAD, SOP, and SAD
* Child and/or parent meets diagnoses (e.g., primary, secondary, tertiary) for any one of the following: pervasive developmental disorders, mental retardation, selective mutism, organic mental disorders, schizophrenia, and other psychotic disorders
* Child and/or parent shows high likelihood and/or serious intent of hurting self or others
* Full-scale IQ score less than 80
* Victim of previously undisclosed abuse requiring investigation or ongoing supervision by the Department of Social Services

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 341 (Actual)
Dates: Start 2008-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinician Severity Rating on the Anxiety Disorders Interview Schedule for Children (ADIS C/P) | Measured at pretreatment, midtreatment, post-treatment, and Year 1 follow up

SECONDARY OUTCOMES:
Child Manifest Anxiety Scale for Children, Revised | Measured at pretreatment, midtreatment, post-treatment, and Year 1 follow up

CONTACTS AND LOCATIONS:
Overall Officials: Wendy K. Silverman, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

REFERENCES:
- [Derived] Patriarca GC, Rey Y, Marin CE, Yeguez CE, Pettit JW, Silverman WK. Parent involvement enhances CBTs for anxiety disorders in Hispanic/Latino youth: Acculturation as a moderator. J Consult Clin Psychol. 2022 Oct;90(10):827-836. doi: 10.1037/ccp0000770. PMID 36355650